CLINICAL TRIAL: NCT06133673
Title: Broad Phenotype Children With Autism in Kent, Surrey, and Sussex: Developing a Self-Report Questionnaire Prioritising Individual Self-Care
Brief Title: KSS Autism: Parameters and Future Care
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sussex Community NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: V2 20/07/2023
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Autism; Autism Spectrum Disorder; Quality of Life
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Schools: Prevalence questionnaire data will be collected from 20 schools.
- Autistic children and young people (CYP): 10 semi-structured qualitative interviews will be conducted with autistics CYP.

SUMMARY:
Referrals for autism assessment have greatly increased in the last few years. This means that waiting times are longer for families, and children and young people are struggling to get the support they need. This also means that the number of autistic children and young people there is assumed to be is not correct. A better understanding of the true number of autistic children and young people is needed so that better support for them can be provided.

This research aims to understand what autism looks like in Kent, Surrey, and Sussex (KSS) to better help autistic children and young people. To do this, schools will be asked about the number of autistic children in their school to better understand the number of children and young people with autism in KSS. Secondly, autistic children and young people will be interviewed to find out about the support they need. The information gathered will help the research team to develop a quality-of-life measure, which can be used by schools to help autistic children and young people get the support they need.

DETAILED DESCRIPTION:
Referrals for autism assessment in the UK have significantly increased in recent years, with mean referral rates doubling between 2015 and 2019. With it taking a year or more to reach a diagnostic conclusion, leaving autistic children and young people unidentified and without access to support they desperately need.

Delays in assessment and diagnosis can be exacerbated in areas of hidden deprivation, including marginalised coastal and cities, as well as rural communities. Delayed diagnosis and complex co-occurring mental health conditions lead to poor lifelong outcomes. With early recognition and diagnosis, early intervention can create more impactful changes in the lives of autistic children.

One area with hidden deprivation is Kent, Surrey and Sussex (KSS), though this area has not been investigated for its prevalence rates. Lack of prevalence investigations across KSS mean few interventions understand local autism changes, and listening to children will tell us about their own lived experience. Current evidence either investigates aspects of autism prevalence using older diagnostic criteria, is comparative looking at co-occurring conditions, or simply reports numbers referred. What is not known are current rates across primary schools, as many studies focus on secondary school transition or experiences.

Initial work by Tebruegge carried out a retrospective investigation only in the Maidstone area of Kent by asking all headteachers to report all children with an established diagnosis of autism. Leekam used KSS children as a Language Impairment comparison group. Department of Health in a broader Kent, East Sussex and South-East London Boroughs investigation reported highest quantiles for prevalence for those diagnosed. Prior work by this research team found that one area of West Sussex has seen autism referrals between 2015-2019 increase annually from 61 to 225 (269% increase). Interviews with Special Educational Needs Coordinators (SENCos) conducted by this research team and the Born in Bradford study suggest that a significant number of children in schools with symptoms of autism are not going through the diagnostic process.

The nationwide Clinical Practice Research Datalink (CPRD) primary care database makes a historical understanding of autism problematic, as codes and diagnostic symptoms change over time. Russell shows autism from 1998 to 2018 involves the use of no less than 16 clinical codes. This makes reference to these codes as difficult, hence our change of view from clinical records to current report from schools. However, children with potential autism or social communication issues are referred by General Practitioners, health visitors, Speech and Language Therapists, school nurses, preschool staff, and schoolteachers. It is unusual to accept referrals from parents directly. Within school-based populations there is relative under-diagnosis amongst children from Reception (4 to 5 Years) to Year 6 (10 to 11 years). Children in the age bracket of 6-8 have symptoms that become more apparent as peers overtake social communication abilities as social interaction and school-based play and communication leap in complexity. This makes their needs more apparent. The referrals continue to increase in the age bracket of 8-11, as the social communication gap continues to widen, especially in girls. With this increase, a better estimate of autism prevalence in the KSS area is needed.

With both referrals and needs of autistic children increasing, other areas of their lives are impacted. Evidence does suggest that having autism can negatively impact autistic children's outcomes in later life, for example, living independently, job employment and retention, having social relationships, experiencing poor mental health and quality-of-life. Despite this, there is limited evidence of a measure of quality of life for autistic children to help with their unmet needs and overall quality-of-life in school.

Mulraney and Coghill reported on the commonly used quality-of-life measures used in children (with ADHD). This includes the Pediatric Quality of Life Inventory (PedsQL) and the Child Health and Illness Profile (CHIP-CE). These measures look at the general functioning of children, such as social, emotional, and physical functioning. Though these questionnaires have been used to look at the quality-of-life in children with ADHD, they do not look at autism, and there is no quality-of-life measure specifically for autistic children. Most studies of quality-of-life of high-functioning autistic children have utilized the PedsQL.

For adults, there is a measure of quality-of-life known as the Autism Quality of Life Measure. The ASQoL is a 9-item measure, designed with autistic people in mind, by autistic people, who participated in the development of the measure. However, it was only designed as an add-on to other QoL measure, the World Health Organisation Quality of Life Measure (WHOQoL), the WHO-BREF and the WHO Disabilities module. Thus, this measure is used in conjunction with other QoL measures, suggesting that there is no standalone quality-of-life measure for autistic people. Also, this measure is used in autistic adults, again suggesting that there is no one single quality-of-life for autistic children.

Given the evidence around outcomes for autistic adults, it seems paramount to intervene early, and give autistic children the ability to have their own say in their needs to improve their quality-of-life. It would be beneficial to have a quality-of-life measure specifically for autistic children to improve their future outcomes. Children's views and suggestions on their own care are therefore vital, yet are rarely gathered, which the research team aim to address by modifying the ASQoL, a validated questionnaire which identifies priorities for Quality of Life and Wellbeing for autistic adults, for autistic children to address their needs in school and help them to advocate for their own support.

ELIGIBILITY:
For the survey, the inclusion criteria are:

- Primary and secondary schools in Kent, Surrey and Sussex

For the CYP interviews, the inclusion criteria are:

* Aged 6-16
* Attends a school in Kent, Surrey and Sussex
* Autism diagnosis

For the survey, the exclusion criteria includes:

* Nurseries
* Higher education schools
* Schools outside of Kent, Surrey and Sussex

For the CYP interviews, the exclusion criteria includes:

* Children outside of 6-16 age range
* Children without autism diagnosis
* Non-verbal children
* Parent/carer unable or unwilling to agree for their child to take part

Ages: 6 Years to 16 Years | Sex: All
Age Groups: Child
Study Population: 20 schools across Kent, Surrey and Sussex (KSS) will take part in completing a questionnaire to ascertain autism prevalence in KSS. 10 children and young people (CYP) will take part in an interview to find out about their needs in school to inform a quality of life questionnaire to be used by CYP and school staff in schools.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-09-18 (Estimated); Study Completion 2024-09-18 (Estimated)

PRIMARY OUTCOMES:
Prevalence questionnaire | 5 minutes
  A 6-item non-validated questionnaire that will be used to ask schools about the number of children on their school roll, the number of children with a diagnosis of autism and also other neurodevelopmental conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie McGrevey, Principal Investigator — Sussex Community NHS FT
Locations (1):
- Sussex Community NHS Foundation Trust, Brighton, United Kingdom